CLINICAL TRIAL: NCT06548399
Title: Bacterial Production of LPC and LPA and Symptoms Generation in Inflammatory Bowel Disease Patients With Chronic Abdominal Pain: a Longitudinal Exploratory Study
Brief Title: Longitudinal Study on Bacterial Production of LPC and LPA in Patients With Inflammatory Bowel Disease
Acronym: Long-IBD
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Premysl Bercik, Professor, McMaster University
Other Study IDs: HiREB-16972
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis
Keywords: longitudinal; IBD; bacteria; LPC; LPA; Chron's disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and urine samples will be collected every day for the week periods 1, 2 and 3. Stool and urine samples will be aliquoted in 2mL sterile tubes in anaerobic (in the case of stool samples) and sterile conditions, for future analysis. Samples will be stored in - 81 freezer located in room 4N30, at McMaster University Medical Centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate whether the gut bacteria in IBD patients cause ongoing abdominal pain, even when the disease is calm. Many inflammatory bowel disease (IBD) patients have this pain, regardless of whether their disease is active or not. This might be linked to an imbalance in gut bacteria. Certain IBD patients with persistent abdominal pain experience increased sensitivity in their gut due to bacteria producing LPC and LPA. Our goal is to explore the connection between bacterial LPC/LPA levels and symptoms in IBD patients with long-lasting abdominal pain. Additionally, we aim to pinpoint the specific bacteria responsible for producing LPC/LPA, which in turn causes chronic abdominal pain in these patients.

DETAILED DESCRIPTION:
The human body is inhabited by a complex community of microbes, collectively referred to as "microbiota". A vast majority of these bacteria are found in the lumen of the gastrontestinal tract (colon, small intestine, stomach and esophagus). Several lines of evidence indicate that changes in microbiota (bacteria) may be involved in the origin of different gastrointestinal diseases, including inflammatory Bowel Disease (IBD), with its two main types: Crohn´s disease and Ulcerative colitis.

Our recent data suggest that the gut bacteria have the capability to produce lysophosphatidylcholine (LPC) and its derivative, lysophosphatidic acid (LPA), small lipid molecules that are were shown previously to be involved in the genesis and maintenance of chronic pain. We found that these molecules are higher in stool of patients with Inflammatory Bowel Disease (IBD), but it is unclear whether 1) they are produced by gut bacteria, and 2) whether their production underlies chronic pain in patients with IBD.

The purpose of our study is to determine whether the gut bacteria produce LPC and LPA and induce chronic abdominal pain, which is common in many patients with IBD, even when their colitis is in remission (absence of overt gut inflammation).

In this exploratory longitudinal study, we will recruit patients with IBD, aged 18-70 years, of both sexes, with a history of moderate to severe chronic abdominal pain (as defined by their gastroenterologist), which persists during remission of colitis (absence of overt inflammation on CT or MRI imaging, and baseline fecal calprotectin <200 μg/g of stool) or while having only mild gut inflammation, defined by either colonoscopy (Endoscopic Mayo score: 0-1 or Simple Endoscopic Score for Crohn's Disease score: 0-10). We will recruit 15 patients with baseline stool LPC >200 μg/mg and LPA >100 μg/mg levels after first assessment in screening visit. Recruitment will take place at McMaster University IBD clinic, currently caring for over 1600 patients with IBD (https://www.mcmasteribd.com).

After study participant meets the eligibility criteria and signs the informed consent, we will collect stool and urine samples and abdominal pain scores for 3 weeks, Monday to Friday each week. Daily stool and urine samples (first stool of the day and morning (overnight) urine) will be collected, and LPC/LPA measured by ELISA. Abdominal pain will be assessed daily with a visual analogue scale (VAS). In addition, clinical symptoms will be evaluated by PROMIS (GI Belly Pain, Diarrhea, Constipation and Bloating) and DASS-21 questionnaires at the end of each week, as they assess symptoms during the preceding 7 days. Dietary intake will be assessed at the beginning of each week by a 3-day food diary. The clinical surveys will be provided online, using RedCap software and secure servers already operational within McMaster.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 70 years of age
* Crohn's disease diagnosis with history of past or current moderate or severe chronic abdominal pain that persist despite colitis being in remission (absence of overt inflammation on CT or MRI imaging, and baseline fecal calprotectin of less than 200 μg/g of stool), or in presence of mild inflammation defined by colonoscopy (Simple Endoscopic Score for Crohn's Disease score: 0-10),
* Ulcerative colitis diagnosis with history of past or current moderate or severe chronic abdominal pain that persist despite colitis being in remission (absence of overt inflammation on CT or MRI imaging, and baseline fecal calprotectin less than 200 μg/g of stool) or in presence of mild inflammation defined by colonoscopy (Endoscopic Mayo score: 0-1)

Exclusion Criteria:

* Current acid anti-secretory and antacid medications
* Antibiotics, antibacterial agents or probiotics, currently, or within the last 8 weeks
* Current pain treatment with opioids or NSAIDs (acetaminophen is permitted)
* Alcohol or drug abuse
* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be a risk or that could interfere with data collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of IBD: Crohn's disease or Ulcerative colitis followed at McMaster University's Gastroenterology Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between daily abdominal pain and stool LPC/LPA levels | From enrolment to the end of data/sample collection period at 3 weeks

SECONDARY OUTCOMES:
Correlation between daily abdominal pain and urine LPC/LPA levels | From enrolment to the end of data/sample collection period at 3 weeks
Correlation between daily abdominal pain and abundance of LPC/LPA producing bacteria in the stool | From enrolment to the end of data/sample collection period at 3 weeks

OTHER OUTCOMES:
Associations between weekly average stool LPC/LPA levels and overall gastrointestinal symptoms, anxiety, depression and stress. | From enrolment to the end of data/sample collection period at 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.